CLINICAL TRIAL: NCT00982176
Title: Anatomo-functional Determinants of Cognitive Impairment After Acute Coronary Syndrome: A Brain MRI and Cerebral Perfusion Scintigraphy Study
Brief Title: Determinants of Cognitive Impairment After Acute Coronary Syndrome
Acronym: COSCA
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Université Victor Segalen Bordeaux 2 (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX2007/31
Record Dates: First submitted 2009-05-12; First posted 2009-09-23 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Coronary Syndrome
Keywords: Anatomo-functional determinants; cognitive impairment; coronary syndrome; brain MRI; cerebral perfusion scintigraphy
MeSH Terms: conditions — Angina, Unstable; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Other: Brain MRI and cerebral perfusion scintigraphy

INTERVENTIONS:
Other: Brain MRI and cerebral perfusion scintigraphy — A standard neuropsychological assessment will be performed by a neuropsychologist. The daily life experience study will be performed. Questions will be asked to the patients by a pocket computer (Palm).
  MRI will be performed on a 3 Tesla research MRI. Two Tc-99m-HMPAO SPECT studies will be performed The second SPECT study will be performed after intravenous injection of acetazolamide.

SUMMARY:
The general purpose of the present pathophysiological study is to investigate the relation between cognitive impairment observed after an acute coronary syndrome and the presence of cerebral anatomo-functional abnormalities. This study will improve the investigators' understanding of the disease and will help in early diagnosis and prevention of vascular dementia in this population.

DETAILED DESCRIPTION:
Cognitive impairment is observed in more than 30% of the patients from 3 to 6 months after an acute coronary syndrome. Executive functions are mainly impaired. Cognition tends to progressively deteriorate during the following years, therefore increasing the risk of vascular dementia. Increased age and low educational level are the main risks factors whereas the risk is not modified by the strategy used to obtain a coronary revascularization. Brain imaging studies have demonstrated a vascular leukoencephalopathy in 50% of the patients with a previous history of ischaemic heart disease. However the link between brain anatomo-functional changes and occurrence of cognitive dysfunction remains largely unknown.

50 patients will be included in this study.

Cognition will be evaluated using a standard neuropsychological assessment (investigating executive function, memory, attention, language and visuo-constructive abilities) and a 7 days experience sampling method which evaluates cognition in daily life. Brain anatomo-functional study will include a brain MRI and two Tc-99m-HMPAO SPECT performed respectively with and without intravenous injection of acetazolamide in order to measure cerebral blood-flow and cerebrovascular reserve capacity.

Prospective exploratory study performed in a cohort of patients admitted for evaluation of their cardio-vascular risk factor 4 ±1 months after an acute coronary syndrome.

Patients will be included 4 ± 1 months after a first episode of acute coronary syndrome. A standard neuropsychological assessment will be performed by a neuropsychologist at inclusion and 6 months later. The daily life experience study will be performed during a period of 7 consecutive days following the inclusion. Questions will be asked to the patients 5 times a day by a pocket computer (Palm). MRI will be performed on a 3 Tesla research MRI. Two Tc-99m-HMPAO SPECT studies will be performed, the first one at inclusion and the second one more than 2 days and less than 15 days after the first. The second SPECT study will be performed after intravenous injection of acetazolamide.

Relationship between cognitive impairment and brain anatomo-functional abnormalities will be investigated using a linear regression model.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Age :30 to 65 years
* First acute coronary syndrome occurred 4 ± 1 months before the inclusion
* Able to understand the use of a pocket computer (palm)
* Able to use a pocket computer (palm)
* Able to give informed consent
* Affiliated to social insurance

Exclusion Criteria:

* Past medical history of stroke
* Diamox® injection contraindication
* Dementia
* History of major depression
* Aphasia
* Severe visual deficiency
* Contra-indication to brain MRI
* Contra-indication to HMPAO
* Contra-indication to Acetazolamide
* Patient under safeguard of justice
* For women, ineffective contraceptive method
* Breast-feeding or Pregnant women

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: a cohort of patients admitted for evaluation of their cardio-vascular risk factor 4 ±1 months after an acute coronary syndrome
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
the extent of white matter vascular lesions (leuko encephalopathy) and impairment in executive functions | Day 0

SECONDARY OUTCOMES:
cognitive parameters and the degree of brain atrophy | at 6 months
cognitive parameters and the number of small deep infarct | after the follow-up (6 months)
cognitive parameters and the basal cerebral blood flow and the cerebrovascular reserve capacity. | after the follow-up (6 months)
impairment in executive functions and the extent of white matter vascular lesions (leuko encephalopathy) | at 6 month (end of follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Igor SIBON, MD, Principal Investigator — University Hospital, Bordeaux
Locations (2):
- France (2):
  - CHU de Bordeaux, Bordeaux
  - Hôpital Cardiologique du Haut-Lévêque (CEPTA), Pessac